## Statistical Analysis Plan

Study Title: Social Media Indoor Tanning Study

NCT03834974

## Statistical Analysis Plan

We summarized recruitment, retention, participation, acceptability, contamination, motivation, belief that a tan is attractive, tanning intentions, outdoor tanning, sun protection behaviors, post engagement, and persuasive impact of posts using descriptive statistics. Means and standard deviations (M[SD]) were presented for variables that were normally distributed, and medians and inter-quartile ranges (IQR) were presented for variables that were not. We compared retention, participation, and acceptability rates to our pre-determined benchmarks of >80% as a metric of feasibility. We compared perceived change in motivation for each target health behavior, intentions to outdoor tan, and number of times tanned outside by condition using Wilcoxon rank sum tests as these variables were not normally distributed. We also compared if participants outdoor tanned at follow-up using a chi-squared test. As this pilot feasibility trial was not sufficiently powered to establish efficacy on the belief that a tan is attractive or sun protection behaviors, we did not compare conditions on these variables. Data analyses were conducted using SAS 9.4 (SAS Institute, Inc, Cary, NC).